CLINICAL TRIAL: NCT02140515
Title: Comparison of Assisted Reproductive Technology (ART) Outcomes Between Two Protocols of Induction of Ovulation by Using Recombinant Luteinizing Hormone (rLH) and Recombinant Follicle Stimulating Hormone (rFSH) in Patients With Hypogonadotropic Hypogonadism
Brief Title: Comparison of Assisted Reproductive Technology (ART) Outcomes Between Two Protocols of Induction of Ovulation in Patients With Hypogonadotropic Hypogonadism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: royan-Emb-018
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2012-08

CONDITIONS: Infertility
Keywords: Gonal-F Luveris Assisted Reproductive Technology Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Infertility | interventions — Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit; follitropin alfa; Luteinizing Hormone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Luveris (Active Comparator): Evaluation the effect of Luveris protocol on Induction of ovulation in Patients with Hypogonadotropic Hypogonadism
  Interventions: Drug: Lutropin alfa
- Gonal-F& Luveris (Active Comparator): Evaluation the effect of Gonal-F& Luveris protocols of Induction of ovulation in Patients with Hypogonadotropic Hypogonadism
  Interventions: Drug: Follitropin alfa and Lutropin alfa

INTERVENTIONS:
Drug: Lutropin alfa — Administration of Gonal-F or recombinant Follicle Stimulating Hormone (rFSH)
  Other Names: Follitropin alfa: Gonal-F or recombinant Follicle Stimulating Hormone (rFSH)
  Arms: Luveris
Drug: Follitropin alfa and Lutropin alfa — Administration of (rFSH) and (rLH)
  Other Names: Follitropin alfa: Gonal-F or recombinant Follicle Stimulating Hormone (rFSH) and; Lutropin alfa: Luveris or Recombinant Luteinizing Hormone (rLH)
  Arms: Gonal-F& Luveris

SUMMARY:
We wanted to compare the Assisted Reproductive Technology (ART) outcomes between two protocols of induction of ovulation in patients with Hypogonadotropic Hypogonadism. In the beginning, all patients receive Recombinant Follicle Stimulating Hormone (Gonal-F) and Recombinant Luteinizing Hormone (Luveris). When at least one follicle reaches 14 mm in diameter, Luveris alone is administered for group A and both drugs Gonal-F and Luveris for group B. Finally Assisted Reproductive Technology (ART) results are compared between the two groups.

DETAILED DESCRIPTION:
In this single blind randomized clinical trial, 90 women with a clinical history of hypogonadotrophic hypogonadism who stopped any treatment with gonadotrophins >1 month before study, with a negative progesterone challenge test, low serum gonadotrophins (Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) less than 5.0 IU/l) and oestradiol (less than 100 pg/ml) and normal serum concentrations of thyroid stimulating hormone (TSH), testosterone and prolactin within 6 months before the start of treatment are studied in the Royan Institute. Other causes of infertility are excluded from the study. All patients receive treatment with recombinant follicle stimulating hormone (Gonal-F) and recombinant luteinizing hormone (Luveris). When at least one follicle reaches 14 mm in diameter, 4mg/day oestradiol is administered and patients are randomly divided into two groups: Luveris alone (intervention group) and continued treatment with both drugs Gonal-F and Luveris (control group). When at least one follicle detects a mean diameter of ≥18 mm and serum estradiol level reaches 500-2000 pg/ml, ovarian stimulation is stopped and injection of 10000 IU Human Chorionic Gonadotrophin (hCG) is administrated.

At the end, the number and size of ovarian follicles, endometrial thickness on the day of injection of Human Chorionic Gonadotrophin (hCG), the number of oocytes retrieved, the number of good quality embryos, chemical and clinical pregnancy rate, fertilization rate and implantation rate will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical history of hypogonadotropic hypogonadism, and laboratory test result comply with diagnosis of hypogonadotropic hypogonadism
* Have discontinued gonadotropins or gonadotropin releasing hormone or estrogen-progesterone replacement therapy at least one month before the study
* Have primary or secondary amenorrhea
* Serum Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) <5.0 IU/l and oestradiol <100 pg/ml before initiation of treatment
* Have a negative progesterone challenge test
* Normal serum concentrations of thyroid stimulating hormone (TSH), prolactin and testosterone within 6 months before the start of study
* Be willing and able to comply with the protocol for the duration of the study
* Have given written informed consent prior to any study related procedure

Exclusion Criteria:

* The other causes of infertility.
* History of ovarian hyper stimulation syndrome
* Abnormal gynecological bleeding of undetermined origin
* Previous or current hormone dependent tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
number of follicles | baseline
  Evaluation thre number follicles before injection of Human Chorionic Gonadotrophin (hCG)
Size of follicle | baseline
  Evaluation the size of follicle before injection of Human Chorionic Gonadotrophin (hCG)
Endometrial thickness | 1day
  Evaluation the endometrial thickness at the day of injection of Human Chorionic Gonadotrophin (hCG)

SECONDARY OUTCOMES:
number of oocytes retrieved | 3 days
  Evaluation the number of oocytes retrieved 34-36 hours after Human Chorionic Gonadotrophin (hCG) injection
Fertilization rate | 2 days
  Evaluation the fertilization rate 2-3 days before the embryo transfer
Biochemical pregnancy rate | 2 weeks
  Evaluation the biochemical pregnancy rate 2 weeks after embryo transfer
Clinical pregnancy rate | 4 weeks
  Evaluation the clinical pregnancy rate 4-6 weeks after embryo transfer
Implantation rate | 4 weeks
  Evaluation the implantation rate 4-6 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — Department of Endocrinology and Female Infertility at Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Seyedeh Masoumeh Moosavi Sadat, MSc, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Centre, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://Royaninstitute.org